CLINICAL TRIAL: NCT00303368
Title: Multicenter Study of Tibial Dysplasia in Neurofibromatosis Type I (NF1) Patients
Brief Title: Neurofibromatosis Type 1 (NF1) and Tibial Dysplasia
Acronym: NF1TD
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Jacques D'Astous, Principal Investigator, Shriners Hospitals for Children
Other Study IDs: 9165
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Neurofibromatosis Type 1; Tibial Dysplasia
Keywords: Neurofibromatosis (NF1); Tibial Dysplasia (TD)
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibromatoses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — If the enrollee's private physician includes surgery in the management of his/her disorder, and if tissue is removed to be discarded, permission is obtained to store the specimen in a tissue repository for future research.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study is a multicenter four-year outcome study of the natural history of tibial dysplasia in patients with NF1 and selected patients without NF1. We will obtain information on the natural history, burden, functional and health status, health-related quality of life, and surgical interventions/outcomes of tibial dysplasia. The project will also establish a Core Facility (NOCF) for tissue samples for future studies.

DETAILED DESCRIPTION:
The three specific aims of this study are:

* Specific Aim 1 - To assess health status and health - related quality of life (HRQL) in 50 children and adolescents with NF1 and tibial dysplasia and in NF1 controls. We hypothesize that children and adolescents with NF1 and tibial dysplasia will experience an additional burden of morbidity due to tibial dysplasia and a downward trajectory of health status and HRQL over time.
* Specific Aim 2 - To assess the long term outcome of current treatment in 100 adult patients diagnosed with NF1 and tibial dysplasia in childhood. We hypothesize that better quality of life and function, in adults with NF1 and tibial dysplasia, are associated with amputation in childhood compared to multiple surgical procedures, the lack of fibular involvement, and fracture later in childhood. We also hypothesize that individuals with NF1 and tibial dysplasia have a higher risk of other bony dysplasias but are at no higher risk of fracture in other bones.
* Specific Aim 3 - To assess the natural history and short-term response to therapy in a cohort of at least 60 children with NF1 and tibial dysplasia and at least 60 children with tibial dysplasia presumably without NF1 prospectively diagnosed during the course of the four-year study period. We hypothesize that NF1 patients with earlier presentation, Crawford Class II A-C, male gender, and the lack of bracing prior to age two are more likely to fracture. We also postulate that individuals with and without NF1 have a similar outcome and response to treatment.

The results of this project will provide a rational basis for future clinical and therapeutic trials.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1:

  * Group 1, NF1 with Tibial Dysplasia, Ages: 3-18
  * Group 2 (control), NF1 without Tibial Dysplasia, Ages 3-18
* Aim 2: NF1 with Tibial Dysplasia, 19+
* Aim 3: Tibial Dysplasia with or without NF1, Ages: birth to 18
* Tissue procurement, any participant undergoing surgery at the tibial site for routine standard of care

Exclusion Criteria:

* Patients without a diagnosis of NF1 or Tibial Dysplasia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with NF1, with or without Tibial Dysplasia, ages 3+ and individuals ages birth through 18 with Tibial Dysplasia, with or without NF1.
Sampling Method: Non-Probability Sample
Enrollment: 395 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John C Carey, MD, MPH, Principal Investigator — University of Utah, Health Science Center
Locations (1):
- Shriners Hospitals for Children, Intermountain Hospital, Salt Lake City, Utah, United States